CLINICAL TRIAL: NCT06729255
Title: A Single Academic Center, Prospective Cohort With Retrospective Loss-of-resistance Comparator, Proof of Concept Study to Evaluate the Safety, Efficacy, and Usability of the EpiZact Device for Parturients Undergoing Epidural Labor Analgesia
Brief Title: A Prospective Cohort Study to Evaluate the Safety, Efficacy, and Usability of the EpiZact Device
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: GuideStar Medical Devices (Unknown)
Responsible Party: Principal Investigator, Brandon M Togioka, Vice Chair of Clinical Research, Anesthesiology and Perioperative Medicine, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00027678
Record Dates: First submitted 2024-12-07; First posted 2024-12-11 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Postdural Puncture Headache; Epidural Analgesia, Obstetric
Keywords: EpiZact; Wet Tap; unintentional dural puncture
MeSH Terms: conditions — Post-Dural Puncture Headache

STUDY DESIGN:
Intervention Model Description: The investigators will perform a prospective cohort with retrospective loss-of-resistance comparator, proof of concept study involving patients undergoing epidural labor analgesia at OHSU University Hospital.
  This is an open-label (unblinded) study.
  The study will involve one arm:
  1) A prospectively enrolled convenience sample of patients that receive epidural labor analgesia with the assistance of the EpiZact device.
  Results will be matched with a sample of patients identified through retrospective chart review that have received standard of care epidural labor analgesia with the loss-of-resistance technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- EpiZact assisted epidural placement (Experimental): All patients enrolled in the study will receive an epidural to treat labor pain with the assistance of the EpiZact device.
  Interventions: Device: EpiZact-assisted epidural placement

INTERVENTIONS:
Device: EpiZact-assisted epidural placement — The standard epidural kit used with the EpiZact device to place a midline epidural using the landmark technique between the L2 and L5 vertebral bodies. The patient's back will be sterilized with a 2% chlorhexidine/70% isopropyl alcohol applicator. The epidural will be placed with a 17-gauge 3.5-inch Tuohy needle. Once the Tuohy needle is appreciated to be engaged in ligament the EpiZact device will be filled with sterile and attached to the Tuohy via a Luer connector. The green button on the EpiZact device will then be pressed to prime the device. The EpiZact device and Tuohy needle will be advanced as a unit in continuous fashion or with intermittent advancement. Upon sensing a loss of resistance, the EpiZact device will provide a visual and tactile signal, halting needle advancement and signaling that the epidural catheter should be threaded through the Tuohy needle.

SUMMARY:
The purpose of the study is to learn more about a new device, the EpiZact Epidural Device, that may be helpful for reducing the likelihood of wet tap when a labor epidural is placed. When epidurals are placed correctly the needle stops just in front of the space in the body that contains cerebrospinal fluid. When the epidural is advanced a short distance further, leakage of cerebrospinal fluid can occur. This is known as a wet tap. A wet tap can result in a severe headache and at times other complications. The goal of this clinical trial is to learn if the use of the EpiZact device prevents wet taps in pregnant women receiving epidurals for relief of labor pain. The main questions this study aims to answer are:

1. What the rate of wet tap with the EpiZact device?
2. What is the rate of failed epidural placement with the EpiZact device?

All patients in the study will receive an epidural with the EpiZact device. The investigators will compare the results with patients not in the study that receive an epidural without the EpiZact device.

DETAILED DESCRIPTION:
The purpose of the study is to learn if use of the EpiZact device decreases the number of wet taps that occur when epidurals are placed. The EpiZact device has a technology that automatically stops the epidural needle when it enters the epidural space. In theory, this should decrease the likelihood of a wet tap. The standard epidural to treat labor pain does not have this capability. The study device may cause fewer wet taps than the standard epidural. All study participants will receive an epidural to treat labor pain with the EpiZact device. Results will be compared with patients receiving epidurals around the same time without the EpiZact device.

If a participant's screening questions show that they can take part in the study, and the participant chooses to be a part of the study, medical records from OHSU or other facilities may be reviewed. Information reviewed may include treatment history, medications, surgeries, allergies, scans, and lab results. The participant will then receive an epidural with the EpiZact device. After the epidural is placed, the participant will be asked a few questions to determine how well the epidural is working and if a complication occurred. The questions are expected to take less than 5 minutes to answer. Participants will also be called 1 week after receiving an epidural to determine if a complication occurred. This call is expected to last less than 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women requesting labor epidural analgesia
* Women pregnant with a single baby (not twins or triplets)

Exclusion Criteria:

* Women requesting not to have a labor epidural
* Height less than 150 cm
* A bleeding disorder, nerve problem, or skin infection that contraindicates receiving an epidural
* A women receiving a combined spinal epidural (CSE) or a dural puncture epidural (DPE)
* A history of spine surgery
* Allergy to local anesthetics (numbing medicine) or skin cleaning solutions
* Decisionally impaired individuals

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with an Unintentional Dural Puncture | 1 week
  Unintentional dural puncture will be a composite outcome diagnosed by any of the following: (1) free flow of cerebrospinal fluid from the Tuohy needle at any time during the epidural technique, (2) requirement of blood patch within one week of neuraxial procedure, or (3) postural headache that worsens with upright posture and improves with supine position diagnosed within one week of neuraxial placement.

SECONDARY OUTCOMES:
Proportion of Participants with Failed Labor Epidural Placement | 2 hours
  Failed epidural placement will be defined as the inability to place a catheter in the epidural place or the need to replace the epidural within 2 hours of insertion. Decision to replace the epidural will be according to standard practice on labor and delivery at OHSU and will typically involve assessment of loss of cold to ice sensation in the lower thoracic and lumbar dermatomes, 50% decrease in labor contraction pain, and new lower extremity paresthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon M Togioka, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to make IPD available to other researchers.